CLINICAL TRIAL: NCT01772381
Title: Dexamethasone in Prevention of Respiratory Morbidity in Elective Caesarean
Brief Title: Dexamethasone in Prevention of Respiratory Morbidity in Elective Caesarean Section in Term Fetus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Noha Rabei, Assistant Professor, Obstetrics and Gynecology, Ain Shams Maternity Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: noharabei
Record Dates: First submitted 2012-12-31; First posted 2013-01-21 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Transient Tachypnea of the Newborn
Keywords: Dexamethasone, term, elective cesarean section
MeSH Terms: conditions — Transient Tachypnea of the Newborn | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexamethasone (Experimental): Dexamethasone, im , 12 mg twice, 12 hrs apart, 48 hrs before elective cesarean section
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Long acting corticosteroid
  Other Names: Decadron

SUMMARY:
Introduction: Babies born at term by elective caesarean section (CS) and before onset of labor are more likely to develop respiratory complications than babies born vaginally. In developing countries resources are scarce and it is difficult to provide expensive treatments as neonatal care.

Aim of the Work: To assess the effect of prophylactic dexamethasone administration before elective cesarean section at term in reducing neonatal respiratory complications.

Patients and methods: 600 women were included in the study and were planned to have elective caesarean section. 300 received dexamethasone 12 mg twice, 12 hours apart 48 hours before delivery. 300 patients were the control group.

The outcomes were: incidence of admission to neonatal intensive care unit (NICU), incidence of transient tachypnea of newborn (TTN), the incidence of respiratory distress syndrome (RDS) and the need for mechanical ventilation.

DETAILED DESCRIPTION:
Dexamethasone which is a long acting corticosteroid can be used prior to elective cesarean section to decrease neonatal respiratory morbidity by enhacing fetal lung maturity.

ELIGIBILITY:
Inclusion Criteria:

* Previous caesarean section
* Complete 37 week calculated from the first day of the last menstrual period.

Exclusion Criteria:

* Obstetric complications such as pre-eclampsia, antepartum hemorrhage or known fetal anomaly.
* Hypertensive patients.
* Chronic disease e.g. diabetes mellitus.
* Known renal disease.
* Pre-operative infection.

Ages: 22 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Special care baby unit | 24 hours
  Special care baby unit admission for babies with respiratory distress

SECONDARY OUTCOMES:
Severity of respiratory distress | 24 hours
  Severity of respiratory distress and the level of care in response

CONTACTS AND LOCATIONS:
Overall Officials: Noha H Rabei, MD, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Sotiriadis A, McGoldrick E, Makrydimas G, Papatheodorou S, Ioannidis JP, Stewart F, Parker R. Antenatal corticosteroids prior to planned caesarean at term for improving neonatal outcomes. Cochrane Database Syst Rev. 2021 Dec 22;12(12):CD006614. doi: 10.1002/14651858.CD006614.pub4. PMID 34935127